CLINICAL TRIAL: NCT05317455
Title: Regulation of Brain Glucose Metabolism in Type 1 Diabetes
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Raimund Herzog, Associate Professor of Medicine, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2000035036
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus, Type 1; Hypoglycemia Unawareness
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Dichloroacetic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): oral solution with flavoring agent, no active drug.
  Interventions: Drug: Dichloroacetate
- Dichloroacetate (Active Comparator): oral solution of dichloroacetate with flavoring agent
  Interventions: Drug: Dichloroacetate

INTERVENTIONS:
Drug: Dichloroacetate — Dichloroacetate has a long safety record of administration to humans with a rare metabolic disorder for over 40 years. It has been given orally to patients with T2DM for up to a week without any problems and other laboratory or significant clinical adverse effects were not noted. It activates mitochondrial PDH flux, a key regulator of glucose oxidation.
  Other Names: DCA

SUMMARY:
This is a prospective randomized placebo-controlled double-blind crossover pilot study determining the effect of dichloroacetate on brain function under clamped hypoglycemia in T1DM.

DETAILED DESCRIPTION:
This study is a prospective randomized placebo-controlled double-blind crossover study designed to address the hypothesis that dichloroacetate has the ability to re-activate brain glucose metabolism under clamped hypoglycemia. The study population is comprised of intensively treated persons with T1D with frequent exposure to hypoglycemia, who have cognitive deficits under hypoglycemia that could be attributed to changes in brain glucose oxidation. The investigators will test the experimental compound DCA in a study that determines whether restoring brain glucose metabolism under hypoglycemia helps maintain cognitive function.

ELIGIBILITY:
Inclusion Criteria:

T1DM subjects with:

* a history of severe hypoglycemia and/or hypoglycemia unawareness or
* a history of severe hypoglycemia with a blood glucose <54 mg/dL, requiring the assistance of another person (with recovery after the administration of oral carbohydrate, intravenous glucose, or glucagon) or
* at least 2 values <54mg/dl during 2 weeks of CGMS testing during the week prior to study.

Exclusion Criteria:

* Age < 18 years or >55 years.
* Body weight >85 kg at screening visit
* BMI > 30 (female) and >30 (male) kg/m2.
* Untreated proliferative retinopathy
* carriers of glutathione transferase Z1 (GSTZ-1) gene polymorphisms that predispose to DCA accumulation and toxicity

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function | 1 day
  Measures of reaction time [in milliseconds] and cognitive testing performance under hypoglycemia [percentage].

SECONDARY OUTCOMES:
Brain glucose metabolism | 1 day
  Measurement of brain glucose metabolism under hypoglycemia.

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Herzog, MD, Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Grouped analysis will be made available after the completion of the study within one year after completion of enrollment at the most.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
  For individual participant data meta-analysis